CLINICAL TRIAL: NCT00971932
Title: Open-label, Single-arm, Multicenter, Phase II Study Investigating Cetuximab in Combination With Chemotherapy in the First-line Treatment of Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) in Japanese Subjects
Brief Title: Study of Cetuximab in Combination With Chemotherapy in Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62241-056
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2012-08-10 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Recurrent and/or metastatic; SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab + Cisplatin/Carboplatin + Fluorouracil (5-FU) (Experimental)
  Interventions: Drug: Cetuximab; Drug: Cisplatin/Carboplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Cetuximab — The initial dose of cetuximab will be 400 milligram per square meter (mg/m^2) as an intravenous (IV) infusion over 120 minutes. Subsequent weekly doses will be 250 mg/m^2 as an IV infusion over 60 minutes.
Drug: Cisplatin/Carboplatin — Subjects will receive 100 mg/m^2 cisplatin as an IV infusion over 60 minutes on day 1 of each 3-week treatment cycle. If subject developed non-hematological toxicities to cisplatin, carboplatin (area under curve 5 [AUC5]) will be administered as an IV infusion over 60 to 120 minutes on Day 1 of each 3-week treatment cycle.
Drug: 5-Fluorouracil — Subjects will receive 1000 mg/m^2 per day 5-FU as a continuous IV infusion over 24 hours from day 1 to day 4 of each 3-week treatment cycle.

SUMMARY:
The primary objective of this trial is to assess the antitumor activity of cetuximab when given in combination with cisplatin + 5-Fluorouracil (5-FU) for the first-line treatment of recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN) in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of SCCHN
2. Confirmed epidermal growth factor receptor (EGFR) expression in tumor tissue by immunohistochemistry (IHC)
3. Expected survival is more than 6 months
4. Presence of at least 1 bidimensionally measurable lesion either by computed tomography (CT) scan or magnetic resonance imaging (MRI)
5. Recurrent and/or metastatic SCCHN not suitable for local therapy
6. Greater than or equal to (>=) 20 years of age
7. Karnofsky performance status (KPS) >= 70% at trial entry
8. Neutrophils: >= 1500 per millimeter^3 (1,500/mm^3); platelet count >= 100,000/mm^3; and hemoglobin >= 9 gram per deciliter (g/dL)
9. Total bilirubin less than or equal to (<=) 2 * upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 3 * ULN
10. Creatinine clearance >60 milliliter per minute (mL/min).Calculated based on formulae such as the Cockroft-Gault formula for creatinine clearance
11. Serum calcium within normal range (If serum albumin < 4.0 g/dL, the following adjusted serum calcium concentration should be within normality: Adjusted serum calcium concentration = actual serum calcium (milligram per deciliter [mg/dL]) - 0.8 * [actual serum albumin (g/dL) - 4]
12. Effective contraception if risk of conception exists (applicable for both male and female subjects)
13. Signed written informed consent
14. Japanese (with Japanese citizenship)

Exclusion Criteria:

1. Nasopharyngeal carcinoma
2. Prior systemic chemotherapy, except if given as part of a multimodal treatment, which was completed more than 6 months prior to trial entry
3. Surgery (excluding prior diagnostic biopsy) or irradiation within 4 weeks before trial entry
4. Pregnancy (absence to be confirmed by serum/urine human chorionic gonadotropin [HCG] test) or breastfeeding
5. Known hypersensitivity or allergic reaction against any of the components of the trial treatment including excipients
6. Uncontrolled diabetes, malignant hypertension (defined as systolic blood pressure >= 180 millimeter of mercury [mmHg] and/or diastolic blood pressure >= 130 mmHg under resting conditions) or liver failure
7. Pulmonary fibrosis, acute lung injury or interstitial pneumonia, or with previous medical history of these states
8. Active infection, (infection requiring IV antibiotics, antibacterial, antifungal, or antiviral agent), including active tuberculosis, or known and declared human immunodeficiency virus (HIV)
9. Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency
10. Current other squamous cell carcinoma (SCC) or previous other malignancy (excluding skin cancer except for melanoma and carcinoma in situ of the cervix or digestive tract) within the last 5 years
11. Intake of any investigational medication within 30 days before trial entry
12. Other concomitant anticancer therapies
13. Documented or symptomatic brain or leptomeningeal metastasis
14. Medical or psychological condition that would not permit the subject to complete the trial or sign informed consent including known drug abuse
15. Previous treatment with monoclonal antibody therapy, other signal transduction inhibitors or EGFR targeting therapy
16. Legal incapacity or limited legal capacity
17. Other protocol-defined exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. Smith, MD, Study Director — Merck Serono Co., Ltd., Japan
Locations (10):
- Japan (10):
  - Research Site, Aichi
  - National Cancer Center East Hospital, Chiba
  - Research Site, Ehime
  - Research Site, Hokkaido
  - Research Site, Kanagawa
  - Tokai University, Kanagawa
  - Research Site, Osaka
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo

REFERENCES:
- [Result] Yoshino T, Hasegawa Y, Takahashi S, Monden N, Homma A, Okami K, Onozawa Y, Fujii M, Taguchi T, de Blas B, Beier F, Tahara M. Platinum-based chemotherapy plus cetuximab for the first-line treatment of Japanese patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck: results of a phase II trial. Jpn J Clin Oncol. 2013 May;43(5):524-31. doi: 10.1093/jjco/hyt034. Epub 2013 Mar 10. PMID 23479384

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU): Participants were administered an initial dose of cetuximab 400 milligram per square meter (mg/m^2) intravenous (IV) infusion over 120 minutes followed by subsequent weekly doses of 250 mg/m^2 IV infusion over 60 minutes along with background chemotherapy consisting of cisplatin 100 mg/m^2 IV infusion over 60 to 120 minutes on day 1 of each 3-week treatment cycle and 5-fluorouracil (5-FU) 1000 mg/m^2 per day as a continuous IV infusion over 24 hours from day 1 to day 4 of each 3-week treatment cycle, for up to 6 cycles in the absence of progressive disease (PD) or unacceptable toxicity. If participant developed non-hematological toxicities to cisplatin, carboplatin (area under curve 5 [AUC5]) was administered as IV infusion over 60 to 120 minutes on Day 1 of each 3-week treatment cycle.
Period: Overall Study
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Started | 33 (Number of participants treated.)
Completed | 26
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Investigator's decision | 2
Not completed — Ongoing | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.20 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) According to Modified World Health Organization (WHO) Criteria
Description: Percentage of participants experiencing a complete response [CR] (complete disappearance of measurable and evaluable disease without new lesions) or partial response [PR] (greater than or equal to 50 percent decrease in the sum of the products of diameters [SOPD] of index lesions compared to the baseline SOPD, with no evidence of PD) confirmed by a subsequent assessment no less than 28 days after criteria for response were first met based on modified WHO criteria as assessed by Independent Review Committee (IRC).
Time Frame: Evaluations performed every 6 weeks until progressive disease (PD) reported between day of first participant treated, until cut-off date, 02 March 2011
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 33
percentage of participants | 36.4 [20.4 to 54.9]

2. Secondary Outcome: Best Overall Response (BOR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Percentage of participants with objective response based assessment of confirmed CR or confirmed PR according to RECIST as assessed by IRC. CR are those that persist on repeat imaging study at least 28 days after initial documentation of response. PR are those with greater than or equal to 30 percent decrease in the SOPD of index lesions compared to the baseline SOPD, with no evidence of PD.
Time Frame: Evaluations performed every 6 weeks until PD reported between day of first participant treated, until cut-off date, 02 March 2011
Population: ITT population included all participants who received at least one dose of the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 33
percentage of participants | 45.5 [28.1 to 63.6]

3. Secondary Outcome: Disease Control Rate
Description: Percentage of participants experiencing a CR (complete disappearance of measurable and evaluable disease without new lesions) or PR (>=50 percent decrease in sum of the products of diameters [SOPD] of index lesions compared to baseline SOPD, with no evidence of PD) confirmed by subsequent assessment no less than 28 days after criteria for response were first met) or stable disease [SD] (neither sufficient decrease to qualify for PR nor sufficient increase to qualify for PD) at least once no less than 42 days after first dose of trial treatment based on modified WHO criteria as assessed by IRC.
Time Frame: as for outcome 2
Population: ITT population included all participants who received at least one dose of the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 33
percentage of participants | 87.9 [71.8 to 96.6]

4. Secondary Outcome: Duration of Response
Description: Duration of response according to modified WHO criteria as assessed by IRC was defined as the time from the first assessment of CR or PR until the date of the first occurrence of PD, or until the date of death when death occurred within 60 days of the last tumor assessment or first administration of trial treatment (whichever was last).
Time Frame: Time from first assessment of CR or PR to PD, death or last tumor assessment, reported between day of first participant treated, until cut-off date, 02 March 2011
Population: Subgroup of participants from the study population with a best overall response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 12
months | 2.8 [2.8 to 5.5]

5. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: The PFS time according to modified WHO criteria as assessed by IRC was defined as duration from first administration of trial treatment until PD (radiological or clinical, if radiological progression is not available) or death due to any cause. Only deaths within 60 days of last tumor assessment are considered. Participants without event are censored on the date of last tumor assessment.
Time Frame: Time from first administration of trial treatment to PD, death or last tumor assessment, reported between day of first participant treated, until cut-off date, 02 March 2011
Population: ITT population included all participants who received at least one dose of the study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 33
months | 4.1 [4.0 to 5.5]

6. Secondary Outcome: Overall Survival (OS) Time
Description: Time from first administration of trial treatment to death. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from first administration of trial treatment or last day known to be alive, reported between day of first participant treated, until cut-off date, 02 March 2011
Population: ITT population included all participants who received at least one dose of the study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 33
months | 12.8 [8.7 to NA] — The upper limit of confidence interval (CI) for the median OS time was not estimated because no further events occurred after estimated median survival time of 12.8 months.

7. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure according to modified WHO criteria as assessed by IRC was defined as the time from first administration of trial treatment until the date of the first occurrence of one of the events defining treatment failure: PD assessed by the investigator, discontinuation of treatment due to PD, discontinuation of treatment due to an adverse event (AE), start of any new anticancer therapy, or withdrawal of consent or death within 60 days of the last tumor assessment or first administration of trial treatment.
Time Frame: Time from first administration of trial treatment to treatment failure or last tumor assessment, reported between day of first participant treated, until cut-off date, 02 March 2011
Population: ITT population included all participants who received at least one dose of the study medication. Here number of participants analyzed "N" is signifying those participants for whom trial treatment failed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Number analyzed (Participants) | 29
months | 4.2 [4.1 to 5.6]

ADVERSE EVENTS:
Time Frame: Baseline until 30 days after last trial treatment.
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU)
Serious Adverse Events (participants affected / at risk) | 12/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU) (N=33)
Intracardiac mass (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Esophageal fistula (Gastrointestinal disorders) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
C-reactive protein increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercreatininemia (Metabolism and nutrition disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (5-FU) (N=33)
Leukopenia (Blood and lymphatic system disorders) | 28
Neutropenia (Blood and lymphatic system disorders) | 27
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Anemia (Blood and lymphatic system disorders) | 16
Lymphopenia (Blood and lymphatic system disorders) | 11
Leukocytosis (Blood and lymphatic system disorders) | 4
Neutrophilia (Blood and lymphatic system disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 23
Acne (Skin and subcutaneous tissue disorders) | 21
Alopecia (Skin and subcutaneous tissue disorders) | 20
Pruritus (Skin and subcutaneous tissue disorders) | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7
Rash generalized (Skin and subcutaneous tissue disorders) | 5
Pruritus generalized (Skin and subcutaneous tissue disorders) | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 5
Skin chapped (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2
Stomatitis (Gastrointestinal disorders) | 26
Nausea (Gastrointestinal disorders) | 23
Constipation (Gastrointestinal disorders) | 22
Diarrhea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 12
Cheilitis (Gastrointestinal disorders) | 9
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Anal hemorrhage (Gastrointestinal disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 30
Hypomagnesemia (Metabolism and nutrition disorders) | 27
Hyponatremia (Metabolism and nutrition disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypochloremia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypercreatininemia (Metabolism and nutrition disorders) | 5
Fatigue (General disorders) | 19
Malaise (General disorders) | 7
Injection site extravasation (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Face edema (General disorders) | 2
Chills (General disorders) | 2
Infusion related reaction (General disorders) | 2
Injection site swelling (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 7
Weight decreased (Investigations) | 16
Hemoglobin decreased (Investigations) | 9
Blood albumin decreased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 6
Protein total decreased (Investigations) | 6
Weight increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 2
Blood urea increased (Investigations) | 2
Paronychia (Infections and infestations) | 19
Nasopharyngitis (Infections and infestations) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dysgeusia (Nervous system disorders) | 11
Headache (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 8
Ventricular extrasystoles (Cardiac disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Nephropathy toxic (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 2
Insomnia (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Ocular hyperemia (Eye disorders) | 2
Orthostatic hypotension (Vascular disorders) | 5
Tinnitus (Ear and labyrinth disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other